CLINICAL TRIAL: NCT04751812
Title: The Use of Venous Cannulation Pain for Evaluation of Pain Sensitivity in an Attempt to Guide Pain Therapy During and Following Anesthesia
Brief Title: Venous Cannulation Pain to Guide Choice of Anesthetic Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Halland (Other)
Collaborators: Lund University (Other)
Responsible Party: Principal Investigator, Anna Persson, MD, PhD, Consultant in Anaesthesia and Intensive Care Medicine, Region Halland
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2020-06178
Record Dates: First submitted 2021-02-05; First posted 2021-02-12 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Pain, Postoperative; Pain Prediction; Laparoscopic Surgery; Venous Cannulation Pain; Anesthesia Opioid Free
Keywords: Postoperative pain; Pain prediction; VCP; Venous Cannulation Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Analgesics, Opioid; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participant will be blinded to allocation arm. The anesthesia nurses, the anesthesiologist and the PACU-nurse will not be blinded to the intervention. The assistant nurse performing the postoperative pain assessments will be blinded to allocation group. Once the assistant nurse has performed the assessment the PACU-nurse will decide on treatment depending on allocation and specific instructions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- High-pain Standard of care (Active Comparator): Patients grading pain associated with venous cannulation >=2.0 allocated to standard treatment.
  Interventions: Procedure: Standard of care
- High-pain Multimodal anesthesia with opioids (Experimental): Patients grading pain associated with venous cannulation >2.0 allocated to extra treatment.
  Interventions: Procedure: High-pain multimodal anesthesia with opioids
- Low-pain Standard of care (Active Comparator): Patients grading pain associated with venous cannulation to <2.0 allocated to standard treatment.
  Interventions: Procedure: Standard of care
- Low-pain opioid-free (Experimental): Patient grading pain associated with venous cannualation to <2.0 allocated to opioid-free anesthesia.
  Interventions: Procedure: Low-pain opioid free

INTERVENTIONS:
Procedure: High-pain multimodal anesthesia with opioids — Paracetamol, Etoricoxib, Oxycodone, Ondansetron po. Betamethasone 4 mg iv.
  Anesthesia:
  As "standard" + bolus esketamine 0.25 mg/kg iv + Clonidine 1 µg/kg i.v.
  Postoperative pain treatment:
  At pain NRS ≥ 4 - 5 mg of oxycodone i.v. Paracetamol will be administered every 6 hours. If above is not sufficient bolus Clonidine 1 µg/kg i.v.
  Other Names: More extensive pain treatment
  Arms: High-pain Multimodal anesthesia with opioids
Procedure: Low-pain opioid free — Paracetamol, Etoricoxib, Ondansetron p.o. Betamethasone 4 mg iv.
  Anesthesia:
  Infusion Dexmedetomidin 0.2 mikrogram/kg/h iv started 5 min before induction Induction: Esketamin 0.1mg/kg + Propofol 1.5-2 mg/kg iv + rocuronium 0.5 mg/kg iv Start of surgery: Esketamin 0.1 mg/kg iv. Maintenance of anesthesia: Sevoflurane Dexmedetomidin inf 0.2 mikrogram/kg/h Esketamin inf 0.1-0.3mg/kg/h and 0.1 mg/kg adjusted after BP and HR 30 min before end of surgery Lidocaine 1 mg/kg iv
  Postoperative pain treatment:
  • Dexmedetomidin (inf 01-0.2 µg/kg/h) 4 hours postoperative
  If pain NRS ≧3 Esketamin 0.1mg/kg iv + Lidocain 0.5 mg/kg iv (max 4 mg/kg /4 h) If pain NRS ≧3 within 30 min after treatment above is given with Esketamin + Lidocain, 2.5 mg Oxycodone iv. is given and may be repeated.
  Other Names: Opioid free anesthesia
  Arms: Low-pain opioid-free
Procedure: Standard of care — Paracetamol, Etoricoxib, Oxycodone, Ondansetron p.o. Betamethasone 4 mg iv.
  Anesthesia:
  Target controlled infusion (TCI) with doses of propofol and remifentanil based on age, weight and height. Oxycodone 0.1 mg/kg 30 minutes before cessation of remifentanil.
  Postoperative care:
  At pain NRS ≥ 4 - 5 mg of oxycodone i.v. Paracetamol will be administered every 6 hours. If above is not sufficient bolus Clonidine 1 µg/kg i.v.
  Arms: High-pain Standard of care; Low-pain Standard of care

SUMMARY:
The investigators have recently shown that pain associated with peripheral venous cannulation can be used to predict the risk of postoperative pain, where patients grading their pain associated with venous cannulation (VCP) above 2.0 VAS units had 3.4 times higher risk of moderate or severe postoperative pain after laparoscopic cholecystectomy and 1.7 times higher risk in a mixed group of patients and surgeries.

The aim of this study is to investigate whether pain sensitivity measurements using VCP can be used to choose anesthesia treatment protocol with the aim to lower acute postoperative pain in those with high risk. In patients with low risk we aim to lower the amount of opioids given.

DETAILED DESCRIPTION:
The investigators will perform a randomized controlled trial randomizing patients to different treatment protocols depending on their pain associated with venous cannulation. There will be two set of instructions for perioperative treatment, one for those grading pain associated with venous cannulation <2.0 (low-pain) and another for those grading VCP ≥2.0 (high-pain).

The low-pain group will be randomized to standard treatment or opioid-free anesthesia. The high-pain group will be randomized to standard treatment or extra in form of additives like esketamine and clonidine.

In the low-pain group the investigators aim for non-inferiority with the gain being avoiding opioids. In the high-pain group the investigators aim for lower post-operative pain.

ELIGIBILITY:
Inclusion Criteria:

* Adults with an American Society of Anesthesiologists (ASA) physical status I or II, undergoing elective laparoscopic surgery at Hallands´ hospital.

Exclusion Criteria:

* Inability to understand information regarding the study. Refusal to give consent. Severe cardiovascular disease. AV-block II. Requirement of additional procedures during surgery, like conversion of laparoscopic to open surgery, incomplete registration of study measurements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Acute postoperative pain | Acute, within 1.5 hours after surgery
  Difference in mean APOP between groups (Opioid free vs Standard of care, Multimodal vs Standard of care). Reported as difference in NRS (numeric rating scale; 0-10 with 0 describing no pain and 10 the worst pain imaginable) with confidence interval (CI).

SECONDARY OUTCOMES:
Proportion of patients with moderate-severe postoperative pain | Acute, 24 hours and 3 months after surgery
  Reported as difference in NRS (numeric rating scale; 0-10 with 0 describing no pain and 10 the worst pain imaginable) with confidence interval (CI).
Association between pain catastrophizing scale and venous cannulation pain | Preoperative measurement
  Correlation between values on the pain catastrophizing scale and venous cannulation pain measured on a visual analog scale (0.0-10.0 with 0.0 describing no pain and 10.0 the worst pain imaginable)
Association between pain catastrophizing and postoperative pain | Acute, within 24 hours after surgery
  Correlation between values on the pain catastrophizing scale and postoperative pain measured on a numeric rating scale (0-10 with 0 describing no pain and 10 the worst pain imaginable)
Association between pain catastrophizing and postoperative pain | At 3 months after surgery
  Correlation between values on the pain catastrophizing scale and postoperative pain measured on a numeric rating scale (0-10 with 0 describing no pain and 10 the worst pain imaginable)
Persistent postoperative pain | At three months after surgery
  Difference in occurence of persistent postoperative pain (assessed via a questionnaire as ocurring or not) comparing the pain sensitive group (VCP >2.0) and pain tolerant group (VCP<2.0).
Difference in persistent pain between groups. | Three months after surgery.
  Difference in mean PPOP between groups (Opioid free vs Standard of care, Multimodal vs Standard of care). Reported as difference in NRS (numeric rating scale; 0-10 with 0 describing no pain and 10 the worst pain imaginable) with confidence interval (CI).
  Multimodal vs Standard of care). Reported as difference in NRS with confidence interval (CI).
Venous cannulation pain for prediction of acute postoperative pain | Acute; within 24 hours
  Difference in mean APOP between pain-sensitive and pain-tolerant groups (SOC VCP≥2,0 vs SOC VCP≤1,9). Reported as difference in NRS (numeric rating scale; 0-10 with 0 describing no pain and 10 the worst pain imaginable) with confidence interval (CI).
Venous cannulation pain for prediction of persistent postoperative pain | Three months after surgery
  Difference in ocurrence of PPOP between pain-sensitive and pain-tolerant groups (SOC VCP≥2,0 vs SOC VCP≤1,9). Reported as difference in NRS (numeric rating scale; 0-10 with 0 describing no pain and 10 the worst pain imaginable) with confidence interval (CI).
Quality of recovery | Acute; within 24 hours
  Difference in Quality of recovery (QoR) after 24 hr between groups (OFA vs SOC, MAO vs SOC)? QoR assessed with the QoR-15 validated questionnaire answered by the patient 24 hours post surgery.

OTHER OUTCOMES:
Proportion of patients with APOP depending on venous cannulation pain | Acute; within 24 hours
  Difference in proportion of patients experiencing moderate to severe APOP (NRS ≥ 4.0) between pain-sensitive and pain-tolerant groups (SOC VCP≥2,0 vs SOC VCP≤1,9)

CONTACTS AND LOCATIONS:
Overall Officials: Anna KM Persson, PhD, MD, Principal Investigator — Region Halland
Locations (1):
- Halland Hospital Halmstad, Halmstad, Halland County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mogianos K, Unden J, Persson A. Effect of individualized anesthesia and analgesia on postoperative pain in patients stratified for pain sensitivity: A study protocol for the PeriOPerative individualization trial randomized controlled trial. Acta Anaesthesiol Scand. 2024 Nov;68(10):1532-1540. doi: 10.1111/aas.14487. Epub 2024 Jun 27. PMID 38937954